CLINICAL TRIAL: NCT06531252
Title: Factors Associated With Perioperative Anxiety Among Patients Undergoing Coronary Angiography or Angioplasty: a Cross-sectional Study
Brief Title: Perioperative Anxiety Among Patients Undergoing Coronary Angiography or Angioplasty
Status: Completed | Type: Observational
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Other Study IDs: 83/GCN-HĐĐĐ
Record Dates: First submitted 2024-07-21; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Anxiety
Keywords: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anxiety is defined as apprehension, tension, or uneasiness that originates from the danger which may be internal or external. Anxiety may manifest with symptoms related to behavior, emotions, and cognition. Anxiety is prevalent in patients before interventional procedures and deteriorates postoperative outcomes, for example, elevated level of postoperative pain, increased infection rate, and high mortality rate.

Coronary artery disease is one of the leading causes of mortality, disability, and workforce loss, resulting from the narrowing or obstruction of one or more branches of the coronary arteries due to the accumulation of atherosclerotic plaques. Coronary angiogram and angioplasty are among the most popular diagnostic and treatment tools available to cardiologists. However, patients and their families often experience anxiety before the procedure due to inadequate psychological preparation.

The majority of research about perioperative anxiety focused on surgery. Magnitude of preoperative anxiety as reported in some studies was in the range of 60-80% in the western population while some researchers showed a wider range, which was 11-80%. However, there is a lack of research reporting the prevalence of anxiety among patients arranged for minimally invasive procedures, especially coronary procedures. To the best of our knowledge, a cross-sectional study conducted in Africa among 267 cardiac patients found that 70.4% of them experienced perioperative anxiety. In contrast, similar studies reported that this figure was 35.0% in Europe and 35.7% in Australia. There was significant variation of anxiety level across countries. As a result, it is unacceptable to extrapolate the magnitude of anxiety in one nation to another with different socio-demographic characteristics, healthcare systems and family support. Moreover anxiety levels before surgery are influenced by various factors such as individual susceptibility, age, gender, prior surgical experiences, education, type and complexity of the surgery, current health condition, and socioeconomic status. Identifying risk factors helps healthcare provider to support psychological services during the preoperative visit so that stress can be reduced. Thus, the aim of this study was to evaluate the extent of preoperative anxiety among Vietnamese patients and explore the factors associated with it within the context of Asian culture.

DETAILED DESCRIPTION:
This is a cross-sectional study conducted at University Medical Center Ho Chi Minh City. The patients were included in our study when patients were more than 18 years old and were able to comprehend Vietnamese language. The patients were excluded from study if the patients were unconscious and not oriented. On the procedural day, when the patients were in waiting room at DSA unit, investigators distributed a self-administer questionnaire to patients who had accepted to participate. The questionnaire is constructed from three parts, namely, demographics, perioperative factors, and the anxiety scale. Investigators employed "The Pre-operative Intrusive Thoughts Inventory (PITI)" as a tool to measure the anxiety scale. PITI 20 comprises twenty questions. This valid and reliable tool has Cronbach's Alpha score of 0.91. The English questionnaire was adapted and translated into the Vietnamese language and back to English. The answers contain 4 response options (4-point Likert scale ranging from "not at all" with 0 points, "some of the time" with 1 point, "often" with 2 points, and "most of the time" with 3 points). 0 and 60 points are the highest and lowest score respectively, the author of the tool reported that patients with 15 or more scores on the PITI-20 scale reliably were classified as high preoperative anxiety while participants who scored less than fifteen were classified as low preoperative anxiety. Section A: Demographic characteristics (8 questions) Section B: perioperative factors (4 questions) Section C: Pre-operative Intrusive Thoughts Inventory (PITI) anxiety scale (20 questions).

Categorical and nominal variables were presented as percentages and continuous variables as means and standard deviations. Noncontinuous variables were compared using the chi-square test and continuous variables using Student's t-test. Independent variables were identified via logistic regression. A two-sided p-value of <0.05 was considered to indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* The patients were included in our study when the patients were more than 18 years old and were able to comprehend Vietnamese language.

Exclusion Criteria:

* The patients were excluded from our study if the patients were unconscious and not oriented

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: On the procedural day, when the patients were in waiting room at DSA unit, investigators distributed a self-administer questionnaire to patients who had accepted to participate
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with perioperative anxiety as assessed by "The Pre-operative Intrusive Thoughts Inventory (PITI)" | 08/2022 - 07/2024
  "The Pre-operative Intrusive Thoughts Inventory (PITI)" was employed. PITI 20, comprises twenty questions.The English questionnaire was adapted and translated into the Vietnamese language and back to English. The answers contain 4 response options (4-point Likert scale ranging from "not at all" with 0 points, "some of the time" with 1 point, "often" with 2 points, and "most of the time" with 3 points). 0 and 60 points are the highest and lowest score respectively, the author of the tool reported that patients with 15 or more scores on the PITI-20 scale reliably were classified as high preoperative anxiety while participants who scored less than fifteen were classified as low preoperative anxiety.
Identify demographic characteristics and perioperative factors related to perioperative anxiety | 08/2022 - 07/2024
  Demographic and perioperative factors are age, gender, marital status, occupation, educational status, average monthly income, locality, living situation, previous hospitalization, previous coronary angiography/angioplasty, pre-procedural anesthesia information, indication-to-procedure duration (hours). Logistic regression analysis was employed to indentify which variables were related to perioperative anxiety (according to PITI 20 score) independently.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinto PR, McIntyre T, Nogueira-Silva C, Almeida A, Araujo-Soares V. Risk factors for persistent postsurgical pain in women undergoing hysterectomy due to benign causes: a prospective predictive study. J Pain. 2012 Nov;13(11):1045-57. doi: 10.1016/j.jpain.2012.07.014. Epub 2012 Oct 12. PMID 23063345
- [Background] Starkweather AR, Witek-Janusek L, Nockels RP, Peterson J, Mathews HL. Immune function, pain, and psychological stress in patients undergoing spinal surgery. Spine (Phila Pa 1976). 2006 Aug 15;31(18):E641-7. doi: 10.1097/01.brs.0000231795.85409.87. PMID 16915080
- [Background] Takagi H, Ando T, Umemoto T; ALICE (All-Literature Investigation of Cardiovascular Evidence) Group. Perioperative depression or anxiety and postoperative mortality in cardiac surgery: a systematic review and meta-analysis. Heart Vessels. 2017 Dec;32(12):1458-1468. doi: 10.1007/s00380-017-1022-3. Epub 2017 Jul 13. PMID 28702898
- [Background] Friede A, O'Carroll PW, Thralls RB, Reid JA. CDC WONDER on the Web. Proc AMIA Annu Fall Symp. 1996:408-12. PMID 8947698
- [Background] Erkilic E, Kesimci E, Soykut C, Doger C, Gumus T, Kanbak O. Factors associated with preoperative anxiety levels of Turkish surgical patients: from a single center in Ankara. Patient Prefer Adherence. 2017 Feb 28;11:291-296. doi: 10.2147/PPA.S127342. eCollection 2017. PMID 28280304
- [Background] Chen SB, Hu H, Gao YS, He HY, Jin DX, Zhang CQ. Prevalence of clinical anxiety, clinical depression and associated risk factors in chinese young and middle-aged patients with osteonecrosis of the femoral head. PLoS One. 2015 Mar 19;10(3):e0120234. doi: 10.1371/journal.pone.0120234. eCollection 2015. PMID 25789850
- [Background] Afrassa N, Nega Kassa R, Girma Legesse T. Preoperative anxiety and its associated factors among patients undergoing cardiac catheterization at saint peter Specialized Hospital and Addis Cardiac Center, Addis Ababa, Ethiopia. International Journal of Africa Nursing Sciences. 2022/01/01/ 2022;17:100430. doi:https://doi.org/10.1016/j.ijans.2022.100430
- [Background] Trotter R, Gallagher R, Donoghue J. Anxiety in patients undergoing percutaneous coronary interventions. Heart Lung. 2011 May-Jun;40(3):185-92. doi: 10.1016/j.hrtlng.2010.05.054. Epub 2010 Aug 17. PMID 20723986
- [Background] Kokalj Palandacic A, Ucman S, Novak Sarotar B, Lainscak M. The manifestation of anxiety in patients undergoing elective coronary angiography. Eur Psychiatry. 2023 Jul 19;66(Suppl 1):S69. doi: 10.1192/j.eurpsy.2023.233. eCollection 2023 Mar.
- [Background] Y.B W, G.L F, H.T Y, A.G H. Prevalence and factors associated with preoperative anxiety among elective surgical patients at University of Gondar Hospital. Gondar, Northwest Ethiopia, 2017. A cross-sectional study. International Journal of Surgery Open. 2018/01/01/ 2018;10:21-29. doi:https://doi.org/10.1016/j.ijso.2017.11.001
- [Background] Crockett JK, Gumley A, Longmate A. The development and validation of the Pre-operative Intrusive Thoughts Inventory (PITI). Anaesthesia. 2007 Jul;62(7):683-9. doi: 10.1111/j.1365-2044.2007.05090.x. PMID 17567344